CLINICAL TRIAL: NCT05345691
Title: A Randomized, Double-Blind, Multicenter, Parallel-Arm Phase 3 Study to Compare the Efficacy, Pharmacodynamics, Safety, and Immunogenicity Between Bmab 1000 and Prolia® in Postmenopausal Women With Osteoporosis
Brief Title: Comparison of Efficacy, Pharmacodynamics, Safety, and Immunogenicity Between Bmab 1000 and Prolia® in Postmenopausal Women With Osteoporosis
Acronym: DEVOTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocon Biologics UK Ltd (Industry)
Responsible Party: Sponsor
Organization: Biocon Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1000-PMO-03-G-02
Record Dates: First submitted 2022-04-12; First posted 2022-04-26 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Postmenopausal Women With Osteoporosis
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind (Patient, Investigator)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bmab 1000 (Experimental)
  Interventions: Biological: Bmab 1000
- Prolia®: (Active Comparator)
  Interventions: Biological: Prolia®

INTERVENTIONS:
Biological: Bmab 1000 — 60 mg administered as a single SC (subcutaneous) injection once every 6 months.
  Arms: Bmab 1000
Biological: Prolia® — 60 mg administered as a single SC injection once every 6 months
  Arms: Prolia®:

SUMMARY:
This is a randomized, double-blind, multicenter, parallel-arm, Phase 3 study to compare the efficacy, PK (Pharmacokinetic), PD (Pharmacodynamic), safety, and immunogenicity of Bmab 1000 and Prolia® in postmenopausal women with osteoporosis

DETAILED DESCRIPTION:
The study will consist of 3 study periods: Screening period; Part 1, double-blind active-controlled period; and Part 2, transition period. In the double-blind active-controlled period, eligible Patients will be randomized in a 1:1 ratio to receive either Bmab 1000 or Prolia®. Prior to dosing At Week 52, patients in Prolia® treatment group will be randomized again in a 1:1 ratio to either continue on Prolia® or be transitioned to Bmab 1000. To maintain the study blinding, the patients in the original Bmab 1000 arm will also go through the re-randomization procedure; however, they will continue to receive Bmab 1000. The interventions (Bmab 1000 or Prolia®) will be administered subcutaneously every 6 months. End-of-study visit will be at Week 78 post randomization (Month 18).

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women, aged ≥55 and <80 years at screening. Postmenopausal is defined as 12 months of spontaneous amenorrhea with serum FSH (follicle-stimulating hormone) levels ≥40 mIU/mL at screening or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
2. Evidence of osteoporosis as assessed by lumbar spine (L1-L4) absolute BMD corresponding to a T-score classification ≤-2.5 and ≥-4.0.
3. At least 3 vertebrae in the L1-L4 region and at least one hip joint are evaluable by DXA at screening.
4. Patients with body weight ≥50 to <90 kg at screening.

Exclusion Criteria:

1. Patients with T-score of <-4.0 at the lumbar spine, total hip, or femoral neck.
2. Known history of previous exposure to denosumab (Prolia®, Xgeva®, or any biosimilar denosumab).
3. For prior or ongoing use of any osteoporosis treatment (other than calcium and vitamin D supplements) following points to be considered for the washout periods prior to the screening visit:

   a. Oral bisphosphonate i. Ineligible if used for 3 or more years cumulatively ii. If used for <3 years, a gap of at least 1 year since the last dose is required at the screening visit b. Dose received any time
4. Systemic glucocorticosteroids
5. Patients with ongoing serious infections
6. Evidence of any of the following per the patient's history, DXA, or X-ray review and/or current disease:

   1. Patient in bed rest for 2 or more weeks during the last 3 months prior to screening
   2. Current hyperthyroidism or hypothyroidism
   3. History and/or current hyperparathyroidism or hypoparathyroidism
   4. Current hypocalcemia or hypercalcemia based on albumin-adjusted serum calcium
   5. Any bone disease including bone metastasis or metabolic disease (except for osteoporosis), eg, osteomalacia or osteogenesis imperfecta, rheumatoid arthritis, Paget's disease, ALP (alkaline phosphatase) elevation (at investigator's discretion), Cushing's disease, clinically significant hyperprolactinemia (at investigator's discretion), fibrous dysplasia, malabsorption syndrome which may interfere with the interpretation of the results
   6. History and/or presence of one severe or 3 or more moderate vertebral fractures
   7. History and/or presence of hip fracture or bilateral hip replacement
   8. Presence of an active healing fracture according to assessment of investigator
   9. History of severe skeletal pain with bisphosphonates which, as per the investigator, is a risk to her participation in the trial
   10. Oral/dental or periodontal conditions:

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 479 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Global Ltd, Granta Park, Great Abington,, Cambridge, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 42 sites across 4 countries, and enrolled 479 subjects
Groups:
- Part 1: Bmab 1000; Part 2: Bmab 1000-Bmab 1000; Part 1: Prolia®; Part 2: Prolia®-Bmab 1000; Part 1: Not Applicable; Part 2: Prolia®-Prolia®: Part 1: Patients were randomly assigned at the baseline/randomization visit (Week 0/Day 1) to receive either Bmab 1000 or Prolia using a 1:1 allocation ratio.
  Part 2: All patients who completed Part 1 underwent the re-randomization process prior to the study drug administration at Week 52. Patients in the Prolia arm were randomly assigned in a 1:1 ratio to receive either Bmab 1000 or Prolia, to obtain data after a single switch in patients who had been treated with Prolia. To maintain the study blinding, the patients in the original Bmab 1000 arm also underwent the re-randomization procedure; however, they continued to receive Bmab 1000 treatment in Part 2
Period: Part 1
Arm/Group | Part 1: Bmab 1000; Part 2: Bmab 1000-Bmab 1000 | Part 1: Prolia®; Part 2: Prolia®-Bmab 1000 | Part 1: Not Applicable; Part 2: Prolia®-Prolia®
Started (Part 1: One patient who was randomized to the Prolia treatment group did not receive any dose as the patient discontinued the study (withdrawal of consent) prior to the first dose administration.) | 238 | 240 | 0
Completed ((Week 52)) | 218 | 208 | 0
Not Completed | 20 | 32 | 0
Period: Part 2
Arm/Group | Part 1: Bmab 1000; Part 2: Bmab 1000-Bmab 1000 | Part 1: Prolia®; Part 2: Prolia®-Bmab 1000 | Part 1: Not Applicable; Part 2: Prolia®-Prolia®
Started (Week 78) | 218 | 104 | 104
Completed | 216 | 103 | 103
Not Completed | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bmab 1000: Bmab 1000: 60 mg administered as a single subcutaneous (SC) injection once every 6 months.
- Total: Total of all reporting groups
Arm/Group | Bmab 1000 | Prolia®: | Total
Number analyzed (Participants) | 238 | 241 | 479
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 88 | 172
  >=65 years | 154 | 153 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (5.55) | 66.5 (5.77) | 66.6 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238 | 241 | 479
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 237 | 241 | 478
  Japanese | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 | 3 | 6
  Europe | 235 | 238 | 473

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Lumbar Spine BMD (Bone Mineral Density)
Description: To demonstrate equivalent efficacy between Bmab 1000 and Prolia® based on percentage change from baseline at Week 52 in lumbar spine BMD
Time Frame: Baseline and Week 52
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Bmab 1000 and Prolia: Bmab 1000: 60 mg administered as a single SC (subcutaneous) injection once every 6 months.
Arm/Group | Bmab 1000 and Prolia | Prolia®
Number analyzed (Participants) | 237 | 235
Percent change | 1.698 (0.5115) | 1.440 (0.5089)

2. Secondary Outcome: AUEC (Area Under the Effect Curve) of the Bone Resorption Marker sCTX (Serum C-terminal Telopeptide of Type 1 Collagen)
Description: To demonstrate pharmacodynamic equivalence between Bmab 1000 and Prolia® based on AUEC of the bone resorption marker sCTX from baseline to week 26
Time Frame: Baseline to Week 26
Population: Modified Full Analysis Set
Measure: Mean (Standard Deviation); unit: day*pg/mL
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 179 | 173
day*pg/mL | 127 (85.2) | 123 (77.3)

3. Secondary Outcome: Percentage Change in Lumbar Spine BMD
Description: To demonstrate equivalent efficacy between Bmab 1000 and Prolia® based on percentage change from baseline at Week 26 in lumbar spine BMD
Time Frame: Baseline and Week 26
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 237 | 235
Percent change | 3.872 (0.7885) | 3.699 (0.7860)

4. Secondary Outcome: Percentage Change in Total Hip BMD by DXA (Dual-energy X-ray Absorptiometry)
Description: To demonstrate equivalent efficacy between Bmab 1000 and Prolia® based on percentage change from baseline, at Week 26 and Week 52 in lumbar spine BMD
Time Frame: Baseline upto week 26
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 237 | 235
Percent change | 1.698 (0.5115) | 1.440 (0.5089)

5. Secondary Outcome: Serum Concentrations of P1NP (Procollagen Type 1 N-terminal Propeptide)
Description: To compare bone turnover between Bmab 1000 and Prolia® based on P1NP after the first dose
Time Frame: Baseline up to Week 52
Population: Modified Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 178 | 177
ng/ml | 69.4 (161) | 42.9 (94)

6. Secondary Outcome: Incidence of TEAEs (Treatment-emergent Adverse Events) up to 6 Months After the Second Dose
Description: To compare safety and tolerability of 2 administrations of Bmab 1000 and Prolia® 6 months apart
Time Frame: Baseline up to Week 78
Measure: Count of Participants; unit: Participants
Groups:
- Bmab 1000-Bmab 1000: (Bmab 1000 in Double-blind Active-controlled Period)
- Bmab 1000 -Prolia; Prolia®:-Prolia: (Prolia in Double-blind Active-controlled Period)
Arm/Group | Bmab 1000-Bmab 1000 | Bmab 1000 -Prolia | Prolia®:-Prolia
Number analyzed (Participants) | 218 | 104 | 104
Participants | 55 | 29 | 27

7. Secondary Outcome: Incidence of ADA (Anti-drug Antibody)
Description: To compare immunogenicity between Bmab 1000 and Prolia®
Time Frame: Week 78 (Transition Period)
Population: Safety Analysis Set for Transition Period
Measure: Count of Participants; unit: Participants
Groups:
- Bmab 1000 (Bmab 1000): (Bmab 1000 in Double-blind Active-controlled)
- Bmab 1000 (Prolia); Prolia (Prolia): (Prolia in Double-blind Active-controlled Period)
Arm/Group | Bmab 1000 (Bmab 1000) | Bmab 1000 (Prolia) | Prolia (Prolia)
Number analyzed (Participants) | 218 | 104 | 104
Participants | 46 | 13 | 14

8. Secondary Outcome: Incidence of ADA (Anti-drug Antibody)
Description: To compare immunogenicity between Bmab 1000 and Prolia®
Time Frame: Baseline up to Week 52 (Double-blind Active-controlled Period)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 238 | 240
Participants | 215 | 205

9. Secondary Outcome: Incidence of NAb (Neutralizing Antibody) up to Week 52
Description: To compare immunogenicity between Bmab 1000 and Prolia®
Time Frame: Baseline up to Week 52 (Double-blind Active-controlled Period)
Measure: Count of Participants; unit: Participants
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 238 | 240
Participants | 7 | 5

10. Secondary Outcome: Percentage Change in Total Hip BMD by DXA (Dual-energy X-ray Absorptiometry)
Description: as for outcome 4
Time Frame: Week 52
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 237 | 235
Percent change | 2.224 (0.5532) | 2.132 (0.5513)

11. Secondary Outcome: Incidence of NAb (Neutralizing Antibody) up to Week 52
Description: To compare immunogenicity between Bmab 1000 and Prolia®
Time Frame: Week 78 (Transition Period)
Population: Safety Analysis Set for Transition Period
Measure: Count of Participants; unit: Participants
Groups:
- Bmab 1000 - Prolia; Prolia - Prolia: (Prolia in Double-blind Active-controlled Period)
Arm/Group | Bmab 1000-Bmab 1000 | Bmab 1000 - Prolia | Prolia - Prolia
Number analyzed (Participants) | 218 | 104 | 104
Participants | 3 | 0 | 0

12. Secondary Outcome: Percentage Change From Baseline in Hip BMD
Description: To demonstrate equivalent efficacy between Bmab 1000 and Prolia® based on percentage change from baseline at Week 78 in Hip BMD
Time Frame: Week 78
Population: Full Analysis Set for Transition Period
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Bmab 1000 - Bmab 1000: (Bmab 1000 in Double-blind Active-controlled Period)
- Prolia - Prolia: (Prolia in Double-blind Active-controlled Period
Arm/Group | Bmab 1000 - Bmab 1000 | Bmab 1000 - Prolia | Prolia - Prolia
Number analyzed (Participants) | 216 | 103 | 103
Percent change | 4.011 (2.7744) | 4.052 (3.4300) | 3.483 (2.6155)

13. Secondary Outcome: Percentage Change From Baseline in Femoral BMD
Description: To demonstrate equivalent efficacy between Bmab 1000 and Prolia® based on percentage change from baseline at Week 78 in Femoral BMD
Time Frame: Week 78
Population: Full Analysis Set for Transition Period
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Bmab 1000- Bmab 1000: (Bmab 1000 in Double-blind Active-controlled Period)
Arm/Group | Bmab 1000- Bmab 1000 | Bmab 1000 - Prolia | Prolia - Prolia
Number analyzed (Participants) | 216 | 103 | 103
Percent change | 3.666 (3.6640) | 3.333 (3.5021) | 2.834 (3.9551)

14. Secondary Outcome: Minimum Concentration (Cmin) of sCTX
Description: To compare minimum Concentration (Cmin) of sCTX between Bmab 1000 and Prolia®
Time Frame: baseline to Week 26
Population: Modified Full Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 236 | 227
pg/mL | 41.5 (18.2) | 41.1 (17.8)

15. Secondary Outcome: Denosumab Concentrations at Weeks 26
Description: Serum Concentrations of Denosumab
Time Frame: Weeks 26
Population: Modified Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 185 | 178
ng/mL | 53.6 (119) | 40.7 (88.1)

16. Secondary Outcome: Denosumab Concentrations at Weeks 52
Description: Serum Concentrations of Denosumab
Time Frame: Weeks 52
Population: Modified Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 178 | 177
ng/mL | 69.4 (161) | 42.9 (94.0)

17. Secondary Outcome: Denosumab Concentrations at Weeks 78
Description: Serum Concentrations of Denosumab
Time Frame: Weeks 78
Population: Modified Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Bmab 1000 - Bmab 1000: (Bmab 1000 in Double-blind Activecontrolled Period)
- Prolia - Prolia: (Prolia in Double-blind Activecontrolled Period)
Arm/Group | Bmab 1000 - Bmab 1000 | Bmab 1000 - Prolia | Prolia - Prolia
Number analyzed (Participants) | 176 | 79 | 83
ng/mL | 87.6 (223) | 72.1 (174) | 66.2 (111)

18. Secondary Outcome: Percentage Change From Baseline in Femoral BMD
Description: To demonstrate equivalent efficacy between Bmab 1000 and Prolia® based on percentage change from baseline at Week 52 in Femoral BMD
Time Frame: Week 52
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bmab 1000 | Prolia®:
Number analyzed (Participants) | 237 | 235
Percent change | 2.138 (0.8042) | 1.767 (0.7999)

ADVERSE EVENTS:
Time Frame: 0- 78 weeks
Description: All Deaths, Serious Adverse Events, and Other Adverse Events were described. For Other adverse Events, a threshold of 2% was used.
  Only one Death was reported during part 1 of the study. Total no. of patients at risk for all-cause mortality is different as compared to the participant at risk for SAEs and other AEs reported throughout the study. Throughout the study is defined as all patients who received Bmab1000 throughout the study or Prolia throughout the study i.e. up to week 78.
Arm/Group | Bmab 1000 | Prolia®:
All-Cause Mortality (participants affected / at risk) | 0/342 | 1/240
Serious Adverse Events (participants affected / at risk) | 15/218 | 2/104
Other Adverse Events (participants affected / at risk) | 144/218 | 72/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bmab 1000 (N=218) | Prolia®: (N=104)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Noninfective mastoiditis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bmab 1000 (N=218) | Prolia®: (N=104)
Bronchitis (Infections and infestations) | 7 (8) | 2 (2)
COVID-19 (Infections and infestations) | 10 (10) | 7 (8)
Cystitis (Infections and infestations) | 3 (4) | 4 (4)
Laryngitis (Infections and infestations) | 5 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 13 (16) | 8 (8)
Pharyngitis (Infections and infestations) | 7 (10) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 18 (21) | 12 (14)
Urinary tract infection (Infections and infestations) | 14 (14) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 5 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 (13) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 4 (5)
Headache (Nervous system disorders) | 11 (12) | 5 (6)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 (7) | 8 (8)
Blood parathyroid hormone increased (Investigations) | 2 (3) | 3 (3)
Hypertension (Vascular disorders) | 7 (7) | 4 (4)
Injection site erythema (General disorders) | 3 (4) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
On Protocol signature page, investigator (PI) declares by signing that "I will not disclose information regarding this clinical investigation or publish results of the investigation without authorization from Biocon Biologics UK Limited."

DOCUMENTS (2):
  • Study Protocol (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT05345691/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT05345691/SAP_001.pdf